CLINICAL TRIAL: NCT01466322
Title: An Open-label, Randomised, Crossover Study to Assess the Relative Bioavailability of Different 2mg Formulations of GSK2018682(S1P1 Agonist) in Healthy Volunteers
Brief Title: A Study to Assess the Relative Bioavailability of Different Formulations of GSK2018682, a Sphingosine-1-phosphate Receptor Subtype 1 Agonist, in Healthy Volunteers.
Acronym: P1A114919
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 114919
Record Dates: First submitted 2011-11-03; First posted 2011-11-07 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Healthy volunteers; GSK2018682; Pharmacokinetics; Relapsing Remitting Multiple Sclerosis; Pharmacodynamics
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral formulations of GSK2018682 (Experimental): Three oral formulations of GSK2018682. A: CD2 Capsule; B: CD3 non-micronised Tablet; C: CD3 micronised Tablet; D: CD3 non-micronised Tablet in fed state
  Interventions: Drug: GSK2018682 CD2 Capsule; GSK2018682 CD3 non-micronised Tablet; GSK2018682 CD3 micronised Tablet; GSK2018682 CD3 non-micronised Tablet in fed state

INTERVENTIONS:
Drug: GSK2018682 CD2 Capsule; GSK2018682 CD3 non-micronised Tablet; GSK2018682 CD3 micronised Tablet; GSK2018682 CD3 non-micronised Tablet in fed state — Four single dosing sessions where each regimen A,B C or D will be administered orally in a randomised, cross-over manner. At each dosing session, pharmacokinetic sampling time-points will be the same.

SUMMARY:
GSK2018682 is a potent and selective agonist for the sphingosine-1- phosphate receptor subtype 1 (S1P1) with the potential to be an effective treatment for multiple sclerosis (MS). The immunomodulatory properties of GSK2018682 are related to functional antagonism of S1P1 on lymphocytes, resulting in sequestration of lymphocytes within the lymphoid organs, rendering them incapable of migrating to sites of inflammation and leading to lymphopenia. Orally administered GSK2018682 is very effective in murine experimental autoimmune encephalomyelitis (EAE), an animal model of human MS. This study will assess the relative bioavailability of different oral formulations of GSK2018682 in healthy volunteers. A tablet formulation is desired for progression into future clinical safety and efficacy studies as the current capsule formulation is not suited to large scale manufacture. The information obtained in this study will help to establish the optimal dosing form for future studies, and also determine the effect of food on the pharmacokinetics of GSK2018682.

DETAILED DESCRIPTION:
BACKGROUND:

Multiple sclerosis (MS) is a debilitating, progressive neurological disease characterized by inflammation of the central nervous system (CNS), resulting in demyelination and axonal damage (for review see [Compston, 2008]). The clinical course for ~85% of MS patients at diagnosis is a relapsing remitting (RRMS) form, characterized by recurrent episodes of neurological dysfunction (relapses) interspersed with longer periods of gradual improvement (remissions). Typical symptoms during RRMS include limb weakness, sensory disturbance and visual impairment. Over time, disability accumulates such that after 10 years approximately half of RRMS patients do not suffer further relapses but show gradual progression of disability, termed secondary progressive (SP) MS [Confavreuax, 2000]. Excess mortality due to MS and quality of life is improving through more rapid and accurate diagnosis combined with better complication management and administration of disease modifying therapies [Bronnum, 2006]. However, more efficacious and better tolerated medicines are needed to relieve the considerable social and economic burden associated with MS.

Sphingosine 1 phosphate (S1P) is an endogenous ligand to a conserved family of five G-protein coupled receptors(S1P receptor subtype 1 -5), with effective concentrations (EC50) ranging from submicromolar to nanomolar levels [Chun, 2002]. Validation for a therapeutic approach targeting S1P receptors in autoimmune disease has been provided by the clinical development of FTY720 in MS (fingolimod; Novartis). GSK2018682 is an agonist at recombinant human S1P1 with some activity at S1P5 receptors but displays no agonist activity towards human S1P2, S1P3 or S1P4 up to a concentration of 10 µM. This selectivity is anticipated to minimise known cardiovascular effects mediated by S1P2/3 subtypes. Orally administered GSK2018682 is very effective in murine experimental autoimmune encephalomyelitis (EAE), an animal model of human MS. GSK2018682 has been reasonably tolerated following single oral doses of 0.6mg to 24mg in an ongoing study (P1A114070) in healthy volunteers

STUDY RATIONALE:

Two Phase I studies (P1A114070 & P1A114347) have been conducted in healthy volunteers using GSK2018682 in capsule formulation. These capsules were produced from a single batch of compound (second drug substance campaign, termed CD2) with a particle size of 15 µm (D90). In order to support further clinical development of GSK2018682, a new batch (CD3) of compound has been synthesized that has a slightly larger particle size (29 µm, D90). In addition, it is intended that longer term studies (Proof of Concept and beyond) will be conducted with a tablet form of the drug. There is also a possibility that obtaining a smaller particle size through micronisation of the CD3 batch (to produce particles with diameters of approximately 3.8 µm, D90) may improve bioavailability; so a tablet made from micronized CD3 GSK2018682 is also being developed. In order to ensure appropriate dose selection for future studies, there is a need to investigate the pharmacokinetic profiles of both new tablet forms of GSK2018682 (manufactured from CD3 campaign) and compare these to the original (CD2) capsule formulation. Therefore, this study will evaluate the relative bioavailability of single doses of each of the 3 different formulations (CD2 capsule, CD3 tablet and CD3 micronized tablet) of GSK2018682 in a cross over, randomized, 4 period, open label design. The fourth treatment arm will be added to examine the effect of food on relative bioavailability of the CD3 tablet formulation. The study will also measure the effects of each dose form of GSK2018682 on total lymphocyte counts.

DOSE RATIONALE:

A 2 mg dose will be used in the study as:

* PK can be well quantified at this dose.
* Significant (in excess of 100%) changes in PK parameters will be detectable.
* PK will be below level of quantification by 7 days after dosing.
* S1P1-mediated PD effects on lymphocytes and heart rate have not been detected.
* There is at least a 2 fold cover to exposures that do have PD effects on lymphocytes and heart rate.
* It is very likely to be a dose used in a future Phase II study (given the predicted accumulation ratio and exposure at steady state).

STUDY DESIGN:

This study will investigate single doses of GSK2018682 in a cohort of 16 healthy male and female (of non-childbearing potential) subjects according to a randomized, open-label, 4 way crossover design. The effect of food on the pharmacokinetics of the CD3 tablet formulation will be explored as it is the most likely to be used in a future Phase II study.

Treatment regimens will include:

* CD2 Capsule
* CD3 non-micronised Tablet
* CD3 micronised Tablet
* CD3 non-micronised Tablet under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters significantly outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with lymphocyte counts outside the normal range should always be excluded from enrollment.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MIU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Male subjects must agree to use one of the protocol-approved contraception methods. This criterion must be followed from the time of the first dose of study medication until the study follow up visit.
* BMI within the range 19 - 29 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 285 ml glass of full strength beer or 425 schooner of light beer or 1 glass (100 ml) of wine or 1 (30 ml) measure of spirits.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Subjects who have asthma.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Subjects with a history of tuberculosis or positive tuberculin (PPD) skin test or a chest X-ray suspicious for tuberculosis, any systemic infection or flu-like symptoms within the last 30 days including fever, cough or other respiratory symptoms, vaccination within the last 30 days, known herpetic flares, history of opportunistic fungal infection (e.g., coccidiomycosis, histoplasmosis, mycosis fungoides, etc.).
* Subjects with a history of, or examination suspicious for, skin cancer(s) including melanoma, basal cell or squamous cell carcinoma.
* Systolic blood pressure less than 95 mmHg or greater than 140 mmHg, or diastolic blood pressure less than or equal to 50 mmHg or greater than or equal to 95 mmHg.
* Symptomatic reduction in blood pressure after orthostatic challenge.
* Subjects with resting heart rate less than 55 beats per minute or greater than 90 beats per minute

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-12-22 (Actual); Primary Completion 2011-02-15 (Actual); Study Completion 2011-02-15 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of different oral formulations of GSK2018682 in healthy volunteers | PK sampling at dosing and at 1, 2, 3, 4, 6, 8, 10, 16, 24, 36, 48, 72, 96, 120, and 144 hr post-dose
  -Peak blood concentration (Cmax); -Time of peak blood concentration (tmax); - Area under the blood concentration-time curve up to the last quantifiable time point (AUC(0-t)) and extrapolated to infinite time (AUC (0-∞)); -Terminal half-life (T½ ); -Apparent oral clearance (CL/F)

SECONDARY OUTCOMES:
To investigate the effect of food on the pharmacokinetic parameters of the CD3 tablet formulation of GSK2018682 | High fat breakfast to be provided within 30 mins prior to dosing
  -Cmax, tmax, AUC (0-∞), T½ and apparent oral clearance
Evaluate the effect of different oral formulations of GSK2018682 on lymphocytes in healthy volunteers | Sampling for absolute lymphocyte count at dosing and at 6 and 24 hr post-dose.
  Reduction from baseline in lymphocyte counts
To investigate the safety and tolerability of different oral formulations of GSK2018682 in healthy volunteers (males and females of non childbearing potential) | AE review: from dosing to follow-up; safety lab parameters: at 48 hr post-dose; Telemetry ECG: dosing to 6 hr post-dose; vital signs: pre-dose,1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 hr post-dose.
  -Adverse event monitoring; -Laboratory parameters (haematology, clinical chemistry, urinalysis); -Telemetry ECG; -Vital signs (systolic and diastolic blood pressure, heart rate, respiratory rate, body temperature)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bronnum-Hansen H, Stenager E, Hansen T, Koch-Henriksen H. Survival and mortality rates among Danes with MS. Int MS J. 2006 May;13(2):66-71. PMID 16635423
- [Background] Chun J, Goetzl EJ, Hla T, Igarashi Y, Lynch KR, Moolenaar W, Pyne S, Tigyi G. International Union of Pharmacology. XXXIV. Lysophospholipid receptor nomenclature. Pharmacol Rev. 2002 Jun;54(2):265-9. doi: 10.1124/pr.54.2.265. PMID 12037142
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] Confavreux C, Vukusic S, Moreau T, Adeleine P. Relapses and progression of disability in multiple sclerosis. N Engl J Med. 2000 Nov 16;343(20):1430-8. doi: 10.1056/NEJM200011163432001. PMID 11078767
- [Background] GlaxoSmithKline Document Number JH2009/00002/01. GSK2018682 Investigator's Brochure.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114919 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114919?search=study&search_terms=114919#rs
- Available data/document: Informed Consent Form: 114919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register